CLINICAL TRIAL: NCT04684303
Title: EuroPainClinicsStudy XI (Cryoablation vs Radiofrequency Ablation of Medial Nerve Branches of Dorsal Roots Crossing Z Joints)
Brief Title: EuroPainClinicsStudy XI (Cryo vs RF MB Z Joints)
Acronym: EPCS XI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Europainclinics z.ú. (Other)
Collaborators: Brno University Hospital (Other); Slovak Academy of Sciences (Other Government); Pavol Jozef Safarik University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03595/2020/OZ-31
Record Dates: First submitted 2020-12-15; First posted 2020-12-24 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Intervention Model Description: Prospective observational clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar medial branch RF neurotomy (Experimental): Procedure lumbar medial branch RF neurotomy By raising the temperature of the tip of the electrode to 85 C for 120 seconds. RF generator. Follow-up: before procedure, 3 months, 6 months, 12 months and 24 months after procedure Repeated cryoablation ablation procedures is allowed (when VAS will be > 4 )
  Interventions: Procedure: Lumbar medial branch radiofrequency ablation neurotomy
- Lumbar medial branch cryoablation (Experimental): Procedure lumbar medial branch cryoablation Decreasing the temperature of the electrode to - 85 C for 120 seconds in two cycles.
  Follow-up: before procedure, 3 months, 6 months, 12 months and 24 months after procedure Repeated cryoablation ablation procedures is allowed (when VAS will be =/> 4 )
  Interventions: Procedure: Lumbar medial branch cryo ablation neurotomy

INTERVENTIONS:
Procedure: Lumbar medial branch radiofrequency ablation neurotomy — Procedure based on positive lumbar Z- joint testing followed by medial branch neurotomy
  Arms: Lumbar medial branch RF neurotomy
Procedure: Lumbar medial branch cryo ablation neurotomy — Procedure based on positive lumbar Z- joint testing followed by medial branch neurotomy
  Arms: Lumbar medial branch cryoablation

SUMMARY:
Determine the efficacy of lumbar medial branch neurotomy by radiofrequency and cryoablation in patients with chronic low back pain

DETAILED DESCRIPTION:
Description of the clinical state:

Facet joint pain encompasses a significant portion of the possible sources of pain in patients with vertebrogenic algic syndrome. A typical symptom caused by facet joint irritation of the medial branch nerve is a back pain with intermittent irregular patchy pain spreading to the legs. The cause of this pain is irritation of the medial branch of the dorsal nerve root which innervates a facet joint. Confirmation of the source of the pain involves local anaesthetic blocks of the medial nerve branches in several adjoining vertebral areas. If this test is positive, then the patient's condition is indicated for radiofrequency ablation or cryoablation of the nerve branches.

Description of interventional procedures:

Patients with chronic low back pain with confirmed zygapophysial joint pain after previous two medial branch nerve blocks with positive results are indicated for radiofrequency medial neurotomy or alternative cryoablation neurotomy. Navigation with probes in both cases is arranged and directed according to fluoroscopic imaging.

ELIGIBILITY:
Inclusion Criteria:dsds

* patients aged between 20 and 80
* positive two medial branch nerve blocks with pain relief over 80% during the first 12hours after nerve block application
* positive patient history for facet joint pain
* patients with chronic low back pain for at least 6 months with back pain and leg pain (VAS >=5)
* those who (only if a signature was obtainable), or whose legal guardian, fully understood the clinical trial details and signed the informed consent form

Exclusion Criteria:

* patients with a history of other spinal diseases (compression fracture, spondylitis, tumor)
* women with positive a pregnancy test before the trial or who planned to become
* pregnant within the following 3 years
* other patients viewed as inappropriate by the staff
* disagreement with participation in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline EuroQoL-5 dimension (EQ-5D) value 6m | 6 months follow-up
  EQ-5D-5L self-care, usual activities, pain/discomfort and anxiety/depression
Change from baseline EuroQoL-5 dimension (EQ-5D) value 12m | 12 months follow-up
  EQ-5D-5L self-care, usual activities, pain/discomfort and anxiety/depression
Change from baseline Visual Analog Pain Scale (VAS) of back pain 6m | 6 months follow-up
  VAS 10 point measurement
Change from baseline Visual Analog Pain Scale (VAS) of back pain 12m | 12 months follow-up
  VAS 10 point measurement
Oswestry disability index (ODI) 6m | 6 months follow-up
  The ODI self-administered questionnaire measuring 0-100 scale
Oswestry disability index (ODI) 12m | 12 months follow-up
  The ODI self-administered questionnaire measuring 0-100 scale

SECONDARY OUTCOMES:
Before procedure drug usage | before procedure
  drug usage
Postprocedural drug usage | 12 months follow-up
  drug usage
Appearance and rate of complications related to procedure | 12 months follow-up
  complications
Dose of radiation exposure | 12 months follow-up
  complications

CONTACTS AND LOCATIONS:
Locations (1):
- EuroPainClinics, Bardejov, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided